CLINICAL TRIAL: NCT05789511
Title: High Resolution Electrogastrography (HR-EGG) Assessment in Medically Refractory Gastroparesis
Brief Title: HR-EGG in Medically Refractory Gastroparesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: Baylor College of Medicine (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Alexander Podboy, MD, Assistant Professor, Department of Medicine, Gastroenterology and Hepatology, University of Virginia
Other Study IDs: 210461
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Gastroparesis; Lung Transplant; Complications
Keywords: Gastroparesis; Post- Lung Transplant
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Medically refractory Non-transplanted gastroparesis: Etiology of gastroparesis deemed on clinical grounds to NOT be secondary to lung transplantation process ( diabetes, post-surgery, idiopathic, neuromuscular etc.)
  Gastroparesis defined as > 10% radiotracer remains in the stomach after 4 hour gastric scintigraphy study.
  Medically refractory is defined as lack of clinical response to trial of diet and lifestyle modifications such as small frequent low fat and low fiber meals and trial or contraindications to prokinetic medications for the treatment of gastroparesis
  Case Cohort: Assessment of HR-EGG comparing controls (non lung transplant induced gastroparesis) vs lung transplant induced gastroparesis
  Investigators will further categorize patients into sub- groups based on HR-EGG phenotypes:, such as High Frequency, Low Frequency, High Amplitude, Low Amplitude, Continuous Symptoms, Sensorimotor Symptoms, Mixed Symptoms and Normal on Day.
  Interventions: Device: High Resolution Electrogastography
- Medically refractory Post Lung transplant gastroparesis: Etiology of gastroparesis deemed on clinical grounds to be secondary to lung transplantation process.
  Gastroparesis defined as > 10% radiotracer remains in the stomach after 4 hour gastric scintigraphy study.
  Medically refractory is defined as lack of clinical response to trial of diet and lifestyle modifications such as small frequent low fat and low fiber meals and trial or contraindications to prokinetic medications for the treatment of gastroparesis
  Case Cohort: Assessment of HR-EGG comparing controls (non lung transplant induced gastroparesis) vs lung transplant induced gastroparesis
  Investigators will further categorize patients into sub- groups based on HR-EGG phenotypes:, such as High Frequency, Low Frequency, High Amplitude, Low Amplitude, Continuous Symptoms, Sensorimotor Symptoms, Mixed Symptoms and Normal on Day.
  Interventions: Device: High Resolution Electrogastography

INTERVENTIONS:
Device: High Resolution Electrogastography — a new generation 64- channel high-resolution electrogastrography recording technology by Alimetry Limited that is able to record and analyze body surface gastric mapping/ HR-EGG
  Other Names: body surface gastric mapping

SUMMARY:
The goal of this observational study is to utilize a novel high resolution electrogastrography device to gauge if identification of gastric dysarrythmias can reliably identify patients that will respond to or will require definitive pyloric interventions such as a G-POEM procedure in patients with medically refractory gastroparesis

Aims:

1. Assess for the presence of gastric dysarrythmias in lung transplantation population as compared to alternative etiologies of gastroparesis
2. Assess if presence or absence of gastric dysarrythmias is predictive of response or need of Gastric -per-oral endoscopic myotomy
3. Assess alterations in gastric dysarrthmias following pyloric interventions including G-POEM.

Patients will undergo two surface body surface gastric mapping via the HR-EGG before and after undergoing a gastric per oral endoscopic myotomy as standard clinical care for the treatment of medically refractory gastroparesis

DETAILED DESCRIPTION:
Gastroparesis is a chronic digestive disorder defined by the symptoms of nausea, vomiting, bloating, and abdominal pain in the setting of objectively delayed gastric emptying without mechanical gastric outlet obstruction. Gastroparesis is frequently identified after lung transplantation with incidence rates as high as 44%. Gastroparesis after lung transplantation is of significant concern as complications directly related to gastroparesis, specifically gastroesophageal reflux and aspiration, have been linked to the development of bronchiolitis obliterans syndrome, the primary cause of graft failure and the main cause of late morbidity and mortality following lung transplantation. Effective long-term therapy for medically refractory post-lung transplant gastroparesis represents a significant therapeutic challenge. Current therapies (such as botulinum toxin injection or surgical pyloromyotomy/bypass) are either limited by inconsistent efficacy or by their invasiveness. However, recent advances in endoscopic tunneling techniques have led to the development of gastric per-oral endoscopic myotomy (G-POEM). Initial reports of this technique for treatment of post-lung transplant gastroparesis are encouraging, with excellent preliminary safety and efficacy data. However, currently there are no clinical, endoscopic, or radiographic parameters that reliably predict which patients will respond to G-POEM. This is likely secondary to the multifactorial pathophysiology of gastroparesis. Secondary to this there is an unmet need to develop a widely deployable screening tool that is i) non-invasive, ii) able to reliably divide gastroparesis into pathophysiologic subgroups and iii) be able to guide effective treatments.

In a similar fashion to that of the brain and heart, waves generated at the stomach's surface propagate to the skin via volume conduction. These voltages can be measured with cutaneous electrodes, via gastric electrophysiology (EGG) noninvasively. However, the EGG has not encountered widespread clinical adoption as the ability to both reliably and consistently differentiate gastrocutaneous spatial dysrhythmias has not been possible. However, a novel 'high-resolution EGG' (HR-EGG), a multi-electrode array of 25 or more electrodes, has been shown to capture slow waves with high spatial resolution and extract meaningful spatial (as opposed to spectral) features, including the instantaneous slow wave direction at any given point in space. This coupled with novel deep convolutional neural network (CNN) frameworks and artifact rejection methods, have been able to reliably capture gastric myoelectricspatial abnormalities that correlate with symptom incidence and severity in gastroparesis patients.

Currently, a new generation of high-resolution electrogastrograms recording technology with 64-channel electrode array is being developed by Alimetry Limited that is able to provide body surface gastric mapping (BSGM). This BSGM is able to provide a more complete understanding of the origin and propagation of human gastric slow-wave activity non-invasively, such as frequency and pattern, in high spatiotemporal detail. The system also includes an App for tracking patient-reported symptoms throughout the test.

Our goal is to utilize this proprietary device to gauge if identification of gastric dysarrythmias can reliably identify patients that will respond to or will require definitive pyloric interventions such as a G-POEM procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >17 years old) with medically refractory gastroparesis

Exclusion Criteria:

* Females who are pregnant or lactating (self-reported)
* History of skin allergies to skin adhesives or hydrogels
* History of extreme sensitivity to cosmetics or lotions
* Fragile skin vulnerable to skin tears
* Damaged epigastric skin (open wounds, rash, inflammation)
* Patients unable to remain in a relaxed reclined position for the test duration
* BMI > 35 obtained via chart review

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung Transplant induced gastroparesis body surface gastric mapping via the HR-EGG will be compared to non-lung transplant induced gastroparesis patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Assess the presence of gastric dysarrythmias in lung transplantation population compared to alternative etiologies of gastroparesis | 2 years
  Investigators will categorize patients into sub- groups based on HR-EGG phenotypes:, such as Low GA-RI, High Frequency, Low Frequency, High Amplitude, Low Amplitude, Continuous Symptoms, Sensorimotor Symptoms, Mixed Symptoms and Normal on Day.

SECONDARY OUTCOMES:
Sub-type the specific bioelectrical abnormalities to assess which patterns are associated with symptoms and abnormal emptying across all subjects | 2 years
Assess if presence or absence of gastric dysarrythmias is predictive of response or need of Gastric -per-oral endoscopic myotomy | 2 years
Assess alterations in gastric dysarrythmias following pyloric interventions including G-POEM | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hooft N, Smith M, Huang J, Bremner R, Walia R. Gastroparesis is common after lung transplantation and may be ameliorated by botulinum toxin-A injection of the pylorus. J Heart Lung Transplant. 2014 Dec;33(12):1314-6. doi: 10.1016/j.healun.2014.08.016. Epub 2014 Sep 6. No abstract available. PMID 25443873
- [Background] Camilleri M, Parkman HP, Shafi MA, Abell TL, Gerson L; American College of Gastroenterology. Clinical guideline: management of gastroparesis. Am J Gastroenterol. 2013 Jan;108(1):18-37; quiz 38. doi: 10.1038/ajg.2012.373. Epub 2012 Nov 13. PMID 23147521
- [Background] Podboy A, Hwang JH, Nguyen LA, Garcia P, Zikos TA, Kamal A, Triadafilopoulos G, Clarke JO. Gastric per-oral endoscopic myotomy: Current status and future directions. World J Gastroenterol. 2019 Jun 7;25(21):2581-2590. doi: 10.3748/wjg.v25.i21.2581. PMID 31210711
- [Background] Nanivadekar AC, Miller DM, Fulton S, Wong L, Ogren J, Chitnis G, McLaughlin B, Zhai S, Fisher LE, Yates BJ, Horn CC. Machine learning prediction of emesis and gastrointestinal state in ferrets. PLoS One. 2019 Oct 18;14(10):e0223279. doi: 10.1371/journal.pone.0223279. eCollection 2019. PMID 31626659
- [Background] Angeli TR, Cheng LK, Du P, Wang TH, Bernard CE, Vannucchi MG, Faussone-Pellegrini MS, Lahr C, Vather R, Windsor JA, Farrugia G, Abell TL, O'Grady G. Loss of Interstitial Cells of Cajal and Patterns of Gastric Dysrhythmia in Patients With Chronic Unexplained Nausea and Vomiting. Gastroenterology. 2015 Jul;149(1):56-66.e5. doi: 10.1053/j.gastro.2015.04.003. Epub 2015 Apr 8. PMID 25863217
- [Background] Berry R, Cheng LK, Du P, Paskaranandavadivel N, Angeli TR, Mayne T, Beban G, O'Grady G. Patterns of Abnormal Gastric Pacemaking After Sleeve Gastrectomy Defined by Laparoscopic High-Resolution Electrical Mapping. Obes Surg. 2017 Aug;27(8):1929-1937. doi: 10.1007/s11695-017-2597-6. PMID 28213666
- [Background] Du P, Calder S, Angeli TR, Sathar S, Paskaranandavadivel N, O'Grady G, Cheng LK. Progress in Mathematical Modeling of Gastrointestinal Slow Wave Abnormalities. Front Physiol. 2018 Jan 15;8:1136. doi: 10.3389/fphys.2017.01136. eCollection 2017. PMID 29379448
- [Background] O'Grady G, Angeli TR, Paskaranandavadivel N, Erickson JC, Wells CI, Gharibans AA, Cheng LK, Du P. Methods for High-Resolution Electrical Mapping in the Gastrointestinal Tract. IEEE Rev Biomed Eng. 2019;12:287-302. doi: 10.1109/RBME.2018.2867555. Epub 2018 Aug 29. PMID 30176605
- [Background] Gharibans AA, Kim S, Kunkel D, Coleman TP. High-Resolution Electrogastrogram: A Novel, Noninvasive Method for Determining Gastric Slow-Wave Direction and Speed. IEEE Trans Biomed Eng. 2017 Apr;64(4):807-815. doi: 10.1109/TBME.2016.2579310. Epub 2016 Jun 9. PMID 27305668
- [Background] Gharibans AA, Smarr BL, Kunkel DC, Kriegsfeld LJ, Mousa HM, Coleman TP. Artifact Rejection Methodology Enables Continuous, Noninvasive Measurement of Gastric Myoelectric Activity in Ambulatory Subjects. Sci Rep. 2018 Mar 22;8(1):5019. doi: 10.1038/s41598-018-23302-9. PMID 29568042
- [Background] Agrusa AS, Gharibans AA, Allegra AA, Kunkel DC, Coleman TP. A Deep Convolutional Neural Network Approach to Classify Normal and Abnormal Gastric Slow Wave Initiation From the High Resolution Electrogastrogram. IEEE Trans Biomed Eng. 2020 Mar;67(3):854-867. doi: 10.1109/TBME.2019.2922235. Epub 2019 Jun 12. PMID 31199249